CLINICAL TRIAL: NCT06975722
Title: A Phase 2b, Multi-national, Multi-center, Randomized, Double-blind, Placebo-controlled, Dose-ranging Study Followed by a Long-term Extension to Evaluate the Efficacy and Safety of SAR442970 in Adult Participants With Moderate to Severe Ulcerative Colitis
Brief Title: A Study to Investigate the Efficacy and Safety of SAR442970 in Adult Participants With Ulcerative Colitis
Acronym: COLOR UC
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ACT18134; 2024-515241-41-00 (EU CTIS Number); U1111-1305-7281 (Other: WHO); ACT18134 (Other: Sanofi)
Record Dates: First submitted 2025-04-28; First posted 2025-05-16 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Ulcerative Colitis
MeSH Terms: conditions — Colitis, Ulcerative

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- SAR442970 Dose Regimen A (Experimental): Participants will receive SAR442970 dose regimen A
  Interventions: Drug: SAR442970
- SAR442970 Dose Regimen B (Experimental): Participants will receive SAR442970 dose regimen B
  Interventions: Drug: SAR442970; Drug: Placebo
- Placebo (Placebo Comparator): Participants will receive SAR442970-matching placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: SAR442970 — Route of administration: Subcutaneous
  Arms: SAR442970 Dose Regimen A; SAR442970 Dose Regimen B
Drug: Placebo — Route of administration: Subcutaneous
  Arms: Placebo; SAR442970 Dose Regimen B

SUMMARY:
This is a phase 2b, randomized, double-blind, 3-arm study for the treatment of Ulcerative Colitis. The primary objective of this study is to assess the efficacy of different doses of SAR442970 compared with placebo in participants with moderate to severe Ulcerative Colitis. The total study duration is up to 168 weeks, with a treatment period of up to 158 weeks including an open-label (OL) long-term extension (LTE) period of up to 104 weeks for eligible participants.

ELIGIBILITY:
Inclusion Criteria:

Participants are eligible to be included in the study only if all of the following criteria apply:

* Male or female participants aged 18 to 75 years inclusive, at the time of signing the informed consent
* Participants who have had clinical evidence of active UC for ≥3 months before screening and confirmed by endoscopy during the screening period
* Must have active moderate-to-severe UC at screening as defined by a modified Mayo Score (mMS) of 5 to 9 (without the Physician Global Assessment (PGA), with a minimum Rectal Bleeding (RB) subscore ≥1, a minimum Stool Frequency (SF) subscore ≥1, mMES ≥2 confirmed by central reader, a minimum sum of all subscores of 5, and a minimum disease extent of 15 cm from the anal verge
* Must have received prior treatment for UC (either "a" or "b" below or combination of both):

  1. History of inadequate response to, loss of response to or intolerance to standard treatment with any of the following compounds: amino-salicylates, corticosteroids, methotrexate, azathioprine, or 6-mercaptopurine, or history of corticosteroid dependence (defined as an inability to successfully taper corticosteroids without recurrence of UC) AND history of no prior exposure to Advanced Therapies (ATs), such as a biologic agent used to treat UC or advanced small molecules used to treat UC
  2. History of inadequate response to, loss of response to or intolerance to treatment with ≥1 approved AT such as a biologic agent used to treat UC or advanced small molecules used to treat UC
* Contraceptive use by men and women should be consistent with local regulations regarding the methods of contraception for those participating in clinical studies

Exclusion Criteria:

* Participants are excluded from the study if any of the following criteria apply:
* Participants with active Crohn's Disease (CD), indeterminate colitis or microscopic colitis
* Participants with fecal sample positive for culture/ova for aerobic pathogens or positive for Clostridium difficile B toxin in stools
* Participant with ostomy or ileoanal pouch, prior colectomy or anticipated colectomy during their participation in the study
* Participants with the following ongoing known complications of UC: fulminant disease, toxic megacolon or colonic dysplasia except for adenoma
* Participants with intestinal failure or short bowel syndrome requiring Total Parenteral Nutrition
* History of recurrent or recent serious infection within 4 weeks of screening, or infection(s) requiring hospitalization or treatment with IV anti-infectives within 30 days prior to baseline, or infections(s) requiring oral anti-infectives within 14 days prior to baseline, except as required as part of an anti-Tuberculosis (TB) regimen
* Known history of or suspected significant current immunosuppression.
* History or solid organ transplant or splenectomy
* History of moderate to severe congestive heart failure (New York Health Association Class III or IV), or recent cerebrovascular accident.
* History of demyelinating disease (including myelitis) or neurologic symptoms suggestive of demyelinating disease
* Participants with a history of malignancy or lymphoproliferative disease other than adequately treated localized carcinoma in situ of the cervix or nonmetastatic squamous cell carcinoma, or nonmetastatic basal cell carcinoma of the skin
* Participants with a diagnosis of inflammatory conditions other than UC (including but not limited to systemic lupus erythematosus, systemic sclerosis, myositis, rheumatoid arthritis, primary biliary cirrhosis, multiple sclerosis, Behcet's disease, sarcoidosis, etc.)
* History of Human Immunodeficiency Virus (HIV) infection or positive HIV serology at Screening
* History of Interstitial Lung Disease
* Participants with any of the following results at Screening:

  * Positive (or indeterminate) Hepatitis B surface antigen (HBs Ag) or,
  * Positive total Hepatitis B core antibody (anti-HBc) confirmed by positive Hepatitis B Virus (HBV) Deoxyribonucleic acid (DNA) or,
  * Positive Hepatitis C Virus (HCV) antibody
* Screening laboratory and other analyses showing abnormal results
* History of any other condition which, in the opinion of the Investigator, would put the participant at risk by participation in the protocol

The above information is not intended to contain all considerations relevant to a participant's potential participation in a clinical trial.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 99 (Estimated)
Dates: Start 2025-07-07 (Actual); Primary Completion 2026-12-17 (Estimated); Study Completion 2029-10-17 (Estimated)

PRIMARY OUTCOMES:
Proportion of participants who achieve clinical remission at the end of Week 16 by modified Mayo Score (mMS) | At Week 16
  Clinical remission is based on modified Mayo subscores. The mMS ranges from 0 to 9 with higher scores indicating greater disease severity.

SECONDARY OUTCOMES:
Proportion of participants who achieve endoscopic improvement at Week 16 | At Week 16
  Endoscopic improvement is defined as a modified Mayo Endoscopic Subscore (mMES) of 0 or 1 (where 1 does not include friability). The mMES ranges from 0 to 3 with higher scores indicating greater disease severity.
Proportion of participants who achieve endoscopic improvement at Week 52 | At Week 52
  Endoscopic improvement is defined as an mMES of 0 or 1 (where 1 does not include friability). The mMES ranges from 0 to 3 with higher scores indicating greater disease severity.
Proportion of participants who achieve endoscopic response at Week 16 | At Week 16
  Endoscopic response is defined as an mMES decrease of at least 1.
Proportion of participants who achieve endoscopic response at Week 52 | At Week 52
  Endoscopic response is defined as an mMES decrease of at least 1.
Proportion of participants who achieve endoscopic remission at Week 16 | At Week 16
  Endoscopic remission is defined as an mMES of 0.
Proportion of participants who achieve endoscopic remission at Week 52 | At Week 52
  Endoscopic remission is defined as an mMES of 0.
Proportion of participants who achieve clinical remission by total Mayo Score (MS) at Week 16 | At Week 16
  Clinical remission is defined as total MS ≤2 with no subscore >1. The total Mayo score (MS) is a composite index designed to measure ulcerative colitis (UC) disease activity and consists of 4 subscores: RB and SF, which are patient-reported subscores, Physician's global assessment (PGA), and endoscopic findings. Individual items are rated 0 to 3, giving the composite score a maximum of 12, with higher scores indicating greater disease severity.
Proportion of participants who achieve clinical remission by total Mayo Score (MS) at Week 52 | At Week 52
  Clinical remission is defined as total MS ≤2 with no subscore >1.
Proportion of participants who achieve clinical response by total MS at Week 16 | At Week 16
  Clinical response by total MS is defined as a decrease from baseline in the total MS of ≥3 points and at least 30% reduction from baseline, and a decrease in the RB subscore of ≥1 or an absolute RB subscore of 0 or 1.
Proportion of participants who achieve clinical response by total MS at Week 52 | At Week 52
  Clinical response by total MS is defined as a decrease from baseline in the total MS of ≥3 points and at least 30% reduction from baseline, and a decrease in the RB subscore of ≥1 or an absolute RB subscore of 0 or 1.
Proportion of participants who achieve clinical response by mMS at Week 16 | At Week 16
  Clinical response by mMS is defined as a decrease from baseline in the mMS of ≥2 points and an improvement of ≥30% from baseline plus a decrease in RB subscore ≥1 or an absolute RB subscore ≤1.
Proportion of participants who achieve clinical response by mMS at Week 52 | At Week 52
  Clinical response by mMS is defined as a decrease from baseline in the mMS of ≥2 points and an improvement of ≥30% from baseline plus a decrease in RB subscore ≥1 or an absolute RB subscore ≤1.
Proportion of participants who achieve clinical remission by mMS at Week 52 | At Week 52
  Clinical remission is defined as an mMS score of 0 to 2, including SF subscore of 0 or 1, RB subscore of 0, and mMES of 0 or 1 (score of 1 does not include friability).
Change from baseline in PRO-2 (Patient Reported Outcome) total score (SF and RB) | From Baseline to Week 16 and up to End of Study (approximately 164 weeks)
  PRO-2 (Patient Reported Outcome) score is defined as the sum of Mayo SF and RB subscores.
Change from baseline in mMS (SF, RB, and mMES) | From Baseline to Week 16 and up to End of Study (approximately 164 weeks)
  Each component of the mMS (SF, RB, and mMES) is scored from 0 to 3. The total mMS ranges from 0 to 9 with higher scores indicating greater disease severity.
Change from baseline in Partial Mayo Score (PMS) (SF, RB, and Physician's Global Assessment [PGA]) | From Baseline to Week 16 and up to End of Study (approximately 164 weeks)
  The Partial Mayo Score (PMS) includes the SF, RB, and PGA components. It ranges from 0 to 9 with higher score indicating highest severity.
Proportion of participants who achieve histological improvement by Original Geboes Score (OGS) to assess inflammation in UC | At Week 16
  Histological improvement is defined as OGS ≤3.1. Original Geboes Score (OGS) is a 6-grade classification system that assesses inflammation severity. Each grade includes subgrades for more specific histological features. Assessment uses the worst area of the biopsy rather than the average. Higher grades indicate greater inflammatory activity in the colon.
Proportion of participants who achieve histological remission by Robarts Histopathology Index (RHI) | At Week 16
  Histological remission is defined as RHI ≤3. The Robarts Histopathology Index (RHI) assesses 4 characteristics of mucosal activity, inflammatory infiltrate, lamina propria neutrophils, neutrophils in epithelium, and erosion or ulceration, all of which are rated on a scale of 0 to 3. Each characteristic is weighted to produce a total score ranging from 0 (no disease activity) to 33 (most severe disease activity).
Proportion of participants who achieve histological remission by OGS to assess inflammation in UC | At Week 16
  Histological remission is defined as OGS <2B.1.
Proportion of participants who achieve Histologic Endoscopic Mucosal Improvement (HEMI) | At Week 16
  HEMI is defined by achievement of modified Mayo endoscopic improvement (mMES of 0 or 1 where 1 does not include friability) and histologic improvement (OGS ≤3.1).
Change from baseline in Inflammatory Bowel Disease Questionnaire (IBDQ) | From Baseline to Week 16
  This captures the patient's experience of inflammatory bowel disease (IBD) on 4 domains of functioning and well-being: bowel and systemic symptoms and emotional and social function. The Inflammatory Bowel Disease Questionnaire (IBDQ) is a 32-item instrument assessing health-related quality of life in IBD patients across four dimensions: bowel symptoms (10 items), systemic symptoms (5 items), emotional function (12 items), and social function (5 items). Each question evaluates experiences over the previous two weeks on a 7-point Likert scale from 1 (worst) to 7 (best). The total score ranges from 32 to 224, with higher scores indicating better quality of life. Both domain-specific and overall scores can be calculated.
Serum SAR442970 concentrations | Up to end of study (approximately 164 weeks)
Incidence of Anti-drug Antibodies (ADAs) | Up to end of study (approximately 164 weeks)
Number (percentage) of participants with any Treatment Emergent Adverse Events (TEAEs) during the Induction and Maintenance treatment periods | From start of induction period to Week 52
Number (percentage) of participants with any TEAEs during the Long-term Extension (LTE) period | From Week 52 (start of LTE period) up to end of the study (approximately 164 weeks)

CONTACTS AND LOCATIONS:
Locations (62):
- United States (21):
  - Investigational Site Number: 8400009, Escondido, California
  - Investigational Site Number: 8400006, Lancaster, California
  - Investigational Site Number: 8400025, Thousand Oaks, California
  - Investigational Site Number: 8400024, Jacksonville, Florida
  - Investigational Site Number: 8400030, Kissimmee, Florida
  - Investigational Site Number: 8400003, Lighthouse PT, Florida
  - Investigational Site Number: 8400001, Miami, Florida
  - Investigational Site Number: 8400011, Miami, Florida
  - Investigational Site Number: 8400010, Palmetto Bay, Florida
  - Investigational Site Number: 8400019, Tampa, Florida
  - Investigational Site Number: 8400018, Marietta, Georgia
  - Investigational Site Number: 8400005, Iowa City, Iowa
  - Investigational Site: 8400017, Boston, Massachusetts
  - Investigational Site Number: 8400012, Wyoming, Michigan
  - Investigational Site Number: 8400014, St Louis, Missouri
  - Investigational Site Number: 8400021, New York, New York
  - Investigational Site Number: 8400029, Queens Village, New York
  - Investigational Site Number: 8400002, Chapel Hill, North Carolina
  - Investigational Site Number: 8400013, Harrisburg, Pennsylvania
  - Investigational Site Number: 8400023, Houston, Texas
  - Investigational Site Number: 8400007, Ogden, Utah
- Investigational Site Number: 0360003, Brisbane, Queensland, Australia
- China (6):
  - Investigative Site: 1560005, Guangzhou, Guangdong
  - Investigative Site: 1560002, Nanjing, Jiangsu
  - Investigative Site: 1560008, Suzhou, Jiangsu
  - Investigative Site: 1560003, Wuxi, Jiangsu
  - Investigational Site Number: 1560001, Hangzhou
  - Investigational Site Number: 1560007, Ningbo
- Investigational Site Number: 2030001, Brno, JM, Czechia
- France (6):
  - Investigational Site Number: 2500002, Lille
  - Investigative Site: 2500006, Nice
  - Investigational Site Number: 2500005, Pierre-Bénite
  - Investigational Site Number: 2500001, Saint-Priest-en-Jarez
  - Investigational Site Number: 2500003, Toulouse
  - Investigational Site Number: 2500004, Vandœuvre-lès-Nancy
- Germany (2):
  - Investigational Site Number: 2760001, Minden, Northwest
  - Investigational Site Number: 2760005, Kiel, Schleswig-Holstein
- Hungary (3):
  - Investigational Site Number: 3480003, Budapest
  - Investigative Site: 3480002, Budapest
  - Investigational Site Number: 3480001, Vác
- Japan (6):
  - Investigational Site Number: 3920002, Kashiwa, Chiba
  - Investigational Site Number: 3920006, Ōita, Oita Prefecture
  - Investigational Site Number: 3920005, Hamamatsu
  - Investigational Site Number: 3920003, Hirosaki
  - Investigational Site Number: 3920001, Morioka
  - Investigational Site Number: 3920004, Nishinomiya
- Investigational Site Number: 4980001, Chisinau, Moldova
- Poland (9):
  - Investigational Site Number: 6160006, Wroclaw, Lower Silesian Voivodeship
  - Investigational Site Number: 6160002, Bydgoszcz
  - Investigational Site Number: 6160009, Chojnice
  - Investigational Site Number: 6160007, Katowice
  - Investigational Site Number: 6160005, Sopot
  - Investigative Site: 6160008, Tychy
  - Investigational Site Number: 6160004, Warsaw
  - Investigational Site Number: 6160003, Warsaw
  - Investigational Site Number: 6160001, Wroclaw
- Spain (2):
  - Investigational Site Number: 7240001, Las Palmas de Gran Canaria
  - Investigational Site Number: 7240002, Madrid
- United Kingdom (4):
  - Investigational Site Number: 8260002, Northwich, CHW
  - Investigational Site Number: 8260003, Bury
  - Investigational Site Number: 8260001, London
  - Investigational Site Number: 8260004, London

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org.

REFERENCES:
- See also: ACT18134 Plain Language Results Summary — https://sanofi.trialsummaries.com/Study/StudyDetails?id=26838&tenant=MT_SNY_9011